CLINICAL TRIAL: NCT05990725
Title: A Phase 3b, Open-label Study to Evaluate the Effectiveness and Safety of Lebrikizumab Treatment in Adults and Adolescents With Moderate-to-Severe Atopic Dermatitis
Brief Title: Effectiveness and Safety of Lebrikizumab Treatment in Adults and Adolescents With Moderate-to-Severe Atopic Dermatitis
Acronym: ADhope
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-17923-33; 2023-505558-16 (EudraCT Number)
Record Dates: First submitted 2023-08-07; First posted 2023-08-14 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: Dermatitis; Skin Diseases
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Dermatitis; Skin Diseases | interventions — lebrikizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lebrikizumab (Experimental): Participants will receive loading doses of lebrikizumab 500 milligrams (mg) subcutaneous (SC) injection at Day 1 and Week 2 followed by lebrikizumab 250 mg SC injection, every two weeks (Q2W) from Week 4 to Week 16. At Week 16, the dosing frequency will be reduced to every 4 weeks (Q4W) and will receive lebrikizumab 250 mg SC injection for up to Week 24, last dose of study medication is administered at Week 20.
  Interventions: Biological: Lebrikizumab

INTERVENTIONS:
Biological: Lebrikizumab — Lebrikizumab solution for injection administered subcutaneously.

SUMMARY:
The main purpose of this study is to evaluate the effectiveness of 24 weeks of lebrikizumab in improving disease severity, signs, and symptoms in adults and adolescents with moderate-to-severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Adults and adolescents (aged >=12 to less than [<] 18 years at the time of informed consent form (ICF)/informed assent form (IAF) signature and weighing >=40 kg) who are candidates for systemic AD therapy.
* Chronic AD that has been present for >=1 year before the Screening visit.
* EASI score >=12 at the Day 1/Baseline Visit.
* IGA score >=3 (moderate) (scale of 0 [clear] to 4 [severe]) at the Baseline visit.
* >=10% BSA of AD involvement at the Day 1/Baseline visit.
* History of inadequate response to treatment with topical medications; or determination that topical treatments are otherwise medically inadvisable.
* Completed electronic diary (eDiary) entries for pruritus and sleep-loss for a minimum of 4 of 7 days before Day 1/Baseline.
* Willing and able to comply with all clinic visits and study-related procedures and questionnaires.
* For women of childbearing potential: agree to remain abstinent (refrain from heterosexual intercourse) or to use a highly effective contraceptive method during the treatment period and for at least 4 weeks or 1 menstrual period after the last dose of lebrikizumab.
* Participant must provide signed ICF. Adolescent participants must also provide separate informed assent to enroll in the study and sign and date either a separate IAF or the ICF signed by the parent/legal guardian (as appropriate based on local regulations and requirements).

Exclusion Criteria:

* Prior treatment at any time with tralokinumab, lebrikizumab, or an oral JAK inhibitor.
* Intention to use any concomitant medication or therapy that is not permitted by this protocol or failure to undergo the required washout period for a particular prohibited medication.
* History of anaphylaxis as defined by the Sampson criteria.
* Uncontrolled chronic disease that might require bursts of oral corticosteroids, example, co-morbid severe uncontrolled asthma (defined by an Asthma Control Questionnaire-5 score >=1.5 or a history of >=2 asthma exacerbations within the last 12 months requiring systemic [oral and/or parenteral] corticosteroid treatment or hospitalisation for >24 hours).
* Occurrence of the following types of infection within 3 months of Screening or develop any of these infections before Day 1/Baseline:

  1. Serious (requiring hospitalisation, and/or IV or equivalent oral antibiotic treatment, as per the Investigator's opinion);
  2. Opportunistic
  3. Chronic (duration of symptoms, signs, and/or treatment of 6 weeks or longer);
  4. Recurring (including, but not limited to herpes simplex, herpes zoster, recurring cellulitis, chronic osteomyelitis).
* Known current or chronic infection with hepatitis B virus.
* Known liver cirrhosis and/or chronic hepatitis of any aetiology.
* Known active endoparasitic infections or at high risk of these infections.
* Known or suspected history of immunosuppression, including history of invasive opportunistic infections (example, tuberculosis, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, and aspergillosis) despite infection resolution: or unusually frequent, recurrent, or prolonged infections, per the Investigator's judgement.
* History of human immunodeficiency virus (HIV) infection or known positive HIV serology.
* Any clinically significant laboratory test results from the chemistry or haematology tests obtained at the Screening visit that would jeopardise the patient's participation in the study, per the Investigator's judgement.
* Presence of skin comorbidities that may interfere with study assessments.
* History of malignancy, including mycosis fungoides, within 5 years before the Screening visit, except completely treated in situ carcinoma of the cervix, completely treated and resolved nonmetastatic squamous or basal cell carcinoma of the skin with no evidence of recurrence in the past 12 weeks.
* Severe concomitant illness(es) that in the Investigator's judgement would adversely affect the participation in the study. Any other medical or psychological condition that in the opinion of the Investigator may suggest a new and/or insufficiently understood disease, may present an unreasonable risk to the study participant because of his/her participation in this clinical trial, may make participation unreliable, or may interfere with study assessments.
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-06-23 (Estimated); Study Completion 2025-06-23 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Eczema Area and Severity Index (EASI) Score Less Than or Equal to (<=) 7 at Week 24 | At Week 24
  The EASI is used to assess the severity and extent of AD; it is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and or extensive disease. The severity of erythema, induration/papulation, excoriation, and lichenification will be assessed by the Investigator or trained designee on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. In addition, the extent of AD involvement in each of the 4 body areas will be assessed as a percentage by body area of head/neck, trunk, upper limbs, and lower limbs, and converted to a score of 0 (0%), 1 (0 to 9%), 2 (10 to 29%), 3 (30 to 49%), 4 (50 to 69%), 5 (70 to 89%) and 6 (90 to 100%).

SECONDARY OUTCOMES:
Percentage of Participants Achieving EASI Score <=7, EASI <=5, and EASI <=3 | Baseline up to Week 24
  The EASI is used to assess the severity and extent of AD; it is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and or extensive disease. The severity of erythema, induration/papulation, excoriation, and lichenification will be assessed by the Investigator or trained designee on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. In addition, the extent of AD involvement in each of the 4 body areas will be assessed as a percentage by body area of head/neck, trunk, upper limbs, and lower limbs, and converted to a score of 0 (0%), 1 (0 to 9%), 2 (10 to 29%), 3 (30 to 49%), 4 (50 to 69%), 5 (70 to 89%) and 6 (90 to 100%).
Percentage of Participants Achieving EASI 75 and EASI 90 | Baseline up to Week 24
  The EASI is used to assess the severity and extent of AD; it is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and or extensive disease. EASI 75 is defined as 75% reduction from baseline in the EASI score. EASI 90 is defined as 90% reduction from baseline in the EASI score.
Percentage of Participants with an Investigator Global Assessment (IGA) Score of 0 or 1 and a Reduction Greater Than or Equal to (>=2) Points | Baseline up to Week 24
  The IGA is an instrument used to globally rate the severity of the participants's AD. It is based on a 5-point scale ranging from 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate) and 4 (severe), and a score is selected using descriptors that best describe the overall appearance of the lesions at a given time point. The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting (minimal, palpable induration and significant induration).
Percentage of Participants Achieving Scoring Atopic Dermatitis (SCORAD) 75 and SCORAD 90 | Baseline up to Week 24
  SCORAD is a validated clinical tool for assessing the extent and intensity of AD. There are 3 components: surface involvement, intensity part and subjective assessment. Surface involvement is assessed as proportion of involved surface area segment by segment by applying the rule of 9s. Intensity part of the SCORAD consists of 6 items: erythema, oedema, oozing/crusting, excoriation, lichenification, and dryness. Each item is graded as follows: none (0), mild (1), moderate (2), or severe (3) (for a maximum of 18 total points). Subjective assessment of itch and of sleeplessness is recorded for each symptom using a VAS, where 0 is no itch (or sleeplessness) and 10 is the worst imaginable itch (or sleeplessness), for maximum possible score of 20. The score ranges from 0 to 103, with higher values indicating a more extensive and/or severe condition. SCORAD 75 is defined as 75% reduction in SCORAD from baseline. SCORAD 90 is defined as 90% reduction in SCORAD from baseline.
Percentage Change From Baseline in Modified Total Lesion Symptom Score (mTLSS) | Baseline up to Week 24
  mTLSS combines an evaluation of hand eczema lesions severity including 6 key signs (erythema, desquamation, lichenification/hyperkeratosis, vesiculae, oedema, fissures) and the intensity of pruritus and pain. The seven features of AD of the hand (erythema, scaling, lichenification/hyperkeratosis, vesiculation, oedema, fissures, pruritus/pain) form the composite scale of mTLSS' strength and each one of them scores from 0 (mild) to 3 (severe). The scores is summed, extending from a base estimation of 0 (no signs or symptoms) to the most extreme of 21 (more serious disease).
Percentage of Participants With Pruritus Numerical Rating Scale (NRS) >=4 at Baseline Achieving >=4-Point Improvement in Pruritus NRS | Baseline up to Week 24
  The Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours, with 0 indicating "No itch," and 10 indicating "Worst itch imaginable. Assessments will be recorded by the participant using an eDiary.
Percentage of Participants Achieving Dermatology Life Quality Index (DLQI) 0-1 | Baseline up to Week 24
  The DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's QoL during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicates 0-1 (no effect on patient's life), 2-5 (small effect on patient's life), 6-10 (moderate effect on patient's life), 11-20 (very large effect on patient's life), 21-30 (extremely large effect on patient's life).
Percentage of Participants With DLQI >=4 at Baseline Achieving >=4-Point Improvement in DLQI | Baseline up to Week 24
  DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's QoL during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. High score is indicative of a poor QoL.
Percentage of Participants Achieving Children Dermatology Life Quality Index (cDLQI) 0-1 | Baseline up to Week 24
  cDLQI is validated from adolescents younger than age of 16 years, which is based on a set of 10 questions different from those of the DLQI. The answers to the questions are generally scored on a 4-point scale from 0=not at all or question unanswered, 1=only a little, 2=quite a lot, 3=very much. cDLQI is calculated by summing the score of each question resulting in 0 to 30. Higher the score, the more impairment of the child's life is experienced.
Percentage of Participants With cDLQI >=6 at Baseline Achieving >=6-Point Improvement in cDLQI | Baseline up to Week 24
  cDLQI is validated from adolescents younger than age of 16 years, which is based on a set of 10 questions different from those of the DLQI. The answers to the questions are generally scored on a 4-point scale from 0=not at all or question unanswered, 1=only a little, 2=quite a lot, 3=very much. cDLQI is calculated by summing the score of each question resulting in 0 to 30. Higher the score, the more impairment of the child's life is experienced.
Percentage of Participants With a Sleep-Loss Scale of >=2 Points at Baseline Who Achieve at least 2-point Reduction Using PRO | Baseline up to Week 24
  Sleep loss will be assessed by all participants using a patient-related outcome (PRO) instrument. Participants (and if applicable, with help of parents/caregiver if required) will rate their sleep on a 5-point Likert scale (with scores ranging from 0 [not at all] to 4 [unable to sleep at all]). Assessments will be recorded by the participant using an eDiary.The baseline Sleep-Loss Scale score will be determined based on the average of daily Sleep-Loss Scale scores during the 7 days immediately before the Day 1 or Baseline visit.
Percentage of Participants With Patient-Oriented Eczema Measure (POEM) >=4 at Baseline Achieving >=4-Point Improvement in POEM | Baseline up to Week 24
  The POEM is a 7-item, validated questionnaire completed by the participant (and, if applicable, with help of parents/caregiver if required) to assess disease symptoms. Participants are asked to respond to questions on skin dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping. All answers carry equal weight, with a total possible score ranging from 0 to 28 (answers scored as: No days = 0; 1-2 days = 1; 3-4 days = 2; 5-6 days = 3; every day = 4. A high score is indicative of a poor quality of life. POEM responses will be captured weekly using an eDiary.
Percentage of Participants With Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Related AEs, AEs Leading to Study Treatment Discontinuation, and Adverse Events of Special Interest (AESIs) | Baseline up to follow-up (Week 28)
  An AE is defined as any untoward medical occurrence in a clinical trial participant, regardless of the administration of the IMP and its causal relationship to it. An AE can therefore be any unfavourable/unintended medical occurrence during the participation in the trial, including deterioration of a pre-existing medical condition, an abnormal value in a laboratory assessment, ECG abnormality, or an abnormal finding in the physical examination. An SAE is an AE, which falls into any of the following categories: death, is life-threatening, requires in-patient hospitalisation or prolongs existing hospitalisation, persistent or significant disability or incapacity, congenital anomaly or birth defect, or any other medically important event that may jeopardise the participant or may require intervention to prevent one of the other above outcomes. The following treatment-emergent AEs are being designated as AESIs: conjunctivitis, herpes simplex or zoster infection and parasitic infections.

CONTACTS AND LOCATIONS:
Locations (33):
- Germany (29):
  - Site 34, Augsburg
  - Site 9, Berlin
  - Site 29, Bonn
  - Site 27, Dresden
  - Site 28, Düsseldorf
  - Site 11, Erlangen
  - Site 37, Frankfurt
  - Site 32, Freiburg im Breisgau
  - Site 5, Göttingen
  - Site 15, Hamburg
  - Site 3, Hamburg
  - Site 8, Hamburg
  - Site 23, Heidelberg
  - Site 1, Kiel
  - Site 19, Langenau
  - Site 10, Lübeck
  - Site 26, Mainz
  - Site 6, Mannheim
  - Site 36, Marburg
  - Site 13, München
  - Site 17, München
  - Site 33, München
  - Site 4, Münster
  - Site 12, Oberhausen
  - Site 22, Oldenburg
  - Site 2, Potsdam
  - Site 30, Regensburg
  - Site 7, Rostock
  - Site 18, Tübingen
- Netherlands (2):
  - Site 35, Bergen op Zoom
  - Site 41, Utrecht
- United Kingdom (2):
  - Site 38, Leeds
  - Site 14, York

IPD SHARING:
Plan to Share IPD: No